CLINICAL TRIAL: NCT04037618
Title: An Open-label, Mass Balance Study to Investigate the Absorption, Metabolism and Excretion of [14C]-EYP001a After a Single Oral Dose to Healthy Male Subjects
Brief Title: Mass Balance Study to Investigate the Absorption, Metabolism and Excretion of [14C]-EYP001a After a Single Oral Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-106
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]-EYP001a (Experimental): [14C]-EYP001a dose A containing 100 μCi radioactivity
  Interventions: Drug: [14C]-EYP001a

INTERVENTIONS:
Drug: [14C]-EYP001a — Oral drinking suspension

SUMMARY:
The study is designed to investigate the absorption, metabolism, and excretion of EYP001a as well as the safety/tolerability of EYP001a following the administration of a single oral dose to healthy male volunteers. The EYP001a dose is administered in a [14C]-labeled form to enable detection and quantitation of dose-related material independent of possible biotransformation.

DETAILED DESCRIPTION:
This is a single site, open-label, mass balance phase 1 study.

Six healthy male subjects will receive a single oral dose A of [14C]-EYP001a containing 100 μCi radioactivity.

* Eligibility is assessed during a screening period of up to 4 weeks.
* Subjects will check into the clinic one day prior to dosing (Day -1) for baseline assessments and to (re-)confirm eligibility.
* The study drug will be administered on Day 1, after an overnight fast of at least 10 hours.
* Blood, urine and fecal samples will be collected up to and including Day 4. If the study discharge criteria are not met on Day 4, blood, urine and fecal samples will be collected in 24- hour intervals until the study discharge criteria are met.
* An End of Study Visit will be planned at Day 14 (+/- 1 Day).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent to participate in this study.
* Healthy and free from clinically significant illness or disease as determined by medical history, physical examination, laboratory and other tests at Screening.
* A body weight of ≥60 kg and a body mass index ranging from 18.0 to 35.0 kg/m2 at Screening.
* Subject must agree to minimize the risk of a female partner becoming pregnant from the dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include abstinence from sexual intercourse, a vasectomy no less than 6 months prior to dosing, barrier contraception or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device (which should be placed at least 1 month before the start of the study), tubal ligation (which took place at least 6 months prior to the start of the study), hormonal contraceptive since at least two months and diaphragm with spermicide. If the subject is a sperm donor, the subject must agree not to donate sperm during the study and until 90 days after the last intake of study drug.
* In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements.

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance.
* History or current clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders.
* History of any major surgery within the last 4 weeks before participation in this study or any bone fracture within the last 2 months.
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders.
* Chronic or relevant acute infections.
* History of allergy/ hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator.
* History of any bleeding disorder including prolonged or habitual bleeding, other hematologic disease or cerebral bleeding (e.g. after a car accident) or commotion cerebri.
* Intake of drugs with a long half-life (>24 hours) within 1 month prior to study drug administration.
* Use of any kind of prescription medication from 14 days prior to the administration of the study drug.
* Use of any kind of over-the-counter products and/or natural health products (including food supplements, herbal supplements, etc.) from 7 days prior to the administration of the study drug.
* Participation in another trial with an investigational drug within 2 months prior to administration of the study drug or during the trial.
* The subject is a smoker or uses other nicotine-containing products.
* Alcohol abuse.
* History of drug abuse.
* Blood donation within 3 months prior to administration or during the trial.
* Any laboratory value outside the reference range, unless considered to lack clinical relevance.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Radioactivity-time profiles in whole blood and plasma | Day 1 to Day 4 or until discharge
Cmax | Day 1 to Day 4 or until discharge
  Maximum observed total radioactivity in plasma and whole blood
tmax | Day 1 to Day 4 or until discharge
  Time from dosing to peak total radioactivity in plasma and whole blood
AUC0-24 | 0 to 24 hours
  Area under the total radioactivity-time curve in plasma and whole blood from time zero to 24 hours
[14C]-metabolic profile and identification of metabolites in plasma | Day 1 to Day 4 or until discharge
[14C]-radioactivity in urine | Day 1 to Day 4 or until discharge
[14C]-metabolic profile and identification of metabolites in urine | Day 1 to Day 4 or until discharge
[14C]-radioactivity in feces | Day 1 to Day 4 or until discharge
[14C]-metabolic profile and identification of metabolites in feces | Day 1 to Day 4 or until discharge

SECONDARY OUTCOMES:
Number of subjects with adverse events | Day 1 to Day 4 or until discharge

CONTACTS AND LOCATIONS:
Overall Officials: C. Voors-Pette, MD, Principal Investigator — QPS Netherlands B.V.
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No